CLINICAL TRIAL: NCT06240988
Title: Effects of Constraint Induced Movement Therapy With and Without Motor Imagery Technique on Upper Limb of Children With Hemiparetic Cerebral Palsy
Brief Title: Effects of CIMT With and Without MIT on Upper Limb of Children With Hemiparetic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0743
Record Dates: First submitted 2023-12-26; First posted 2024-02-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: MCIMT, Motor Imagery Technique, Hemiparetic CP, RCT
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be Randomized Controlled Trial in which non probability convenient sampling technique will be used. two groups of 6 to 14 years of age will be formed in which participants will be randomly divided. Group A will be given Modified CIMT and the other group B will receive motor imagery technique on upper limb in hemiparetic CP.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Constraint Induced Movement Therapy (Experimental): Group that will be provided with Modified Constraint Induced Movement Therapy. A protocol of 10 minutes of MCIMT therapy will be given including constraints.
  Interventions: Device: Modified Constraint Induced Movement Therapy
- Motor Imagery Technique (Experimental): Group that will be provided with Motor Imagery Technique by grasping an object and placing it into a container, or in imagining to perform the same action.
  Interventions: Other: Motor Imagery Technique

INTERVENTIONS:
Device: Modified Constraint Induced Movement Therapy — Modified Constraint Induced Movement Therapy
  Arms: Modified Constraint Induced Movement Therapy
Other: Motor Imagery Technique — Motor Imagery Technique
  Arms: Motor Imagery Technique

SUMMARY:
Cerebral Palsy (CP) is a major cause of motor disability in children. Among these CP children, approximately one third have hemiparetic cerebral palsy. Hemiparetic cerebral palsy is more impairment of one side of the body as a result of non-progressive disturbances in premature brain.To determine the effects of implementing a practice period of modified constraint induced movement therapy in a virtual environment on hand function in chidren with hemiparetic cerebral palsy.

DETAILED DESCRIPTION:
To determine the effects of implementing a practice period of modified constraint induced movement therapy in a virtual environment on hand function in chidren with hemiparetic cerebral palsy.The term Modified constraint-induced movement therapy is a form of rehabilitation therapy that limits the less paretic side, and through repeated and concentrated training improve the upper limb function of the paretic side. Motor imagery is a cognitive process in which a subject imagines that he or she performs a movement without actually performing the movement and without even tensing the muscles. Modified Constraint induced movement therapy can be utilized in both the lower and upper extremities with the motor imagery technique for psychological or occupational therapy and in affecting which one is better for speedy recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 14 years were included.
* Diagnosed of hemiparetic cerebral palsy and typically developing controls.
* Both gender is included i-e, male and female.
* Children included having motor impairments of upper limb.
* All children had normal or corrected vision and the ability to discriminate between right and left.

Exclusion Criteria:

* History of neurosensory and neuropsychiatric impairments.
* Presence of contractures in the affected upper limb.
* Surgery in the previous six months.
* Uncontrolled epilepsy

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
QUEST (Quality of Upper Extremity Skills Test) | 8 weeks
  Item The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. The purpose of the QUEST is to evaluate quality of upper extremity function in four domains: dissociated movement,grasp,protective extension, and weight bearing. Scores of 1 or 2, determined by quality of assessed position or movement; 1 if movement quality is not achieved, 2 if movement quality is achieved. Item scores are summed; formulas are used to calculate percentages for each domain. Domain percentages are summed and divided by number of domains to obtain total score. Minimum score = 0, Maximum score = 100.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | 8 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations. Clients are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Score each hand separately. Higher scores are indicative of better manual dexterity. During the performance of the BBT, the evaluator should be aware of whether the client's fingertips are crossing the partition. Blocks should be counted only when this condition is respected. Furthermore, if two blocks are transferred at once, only one block will be counted. Blocks that fall outside the box, after trespassing the partition, even if they don't make it to the other compartment, should be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Khansa Khalid, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humphreys P, Whiting S, Pham B. Hemiparetic cerebral palsy: clinical pattern and imaging in prediction of outcome. Can J Neurol Sci. 2000 Aug;27(3):210-9. PMID 10975533
- [Background] Steenbergen B, Gordon AM. Activity limitation in hemiplegic cerebral palsy: evidence for disorders in motor planning. Dev Med Child Neurol. 2006 Sep;48(9):780-3. doi: 10.1017/S0012162206001666. PMID 16904028